CLINICAL TRIAL: NCT03253341
Title: Prescribing Smart Aging: Integrating Health Systems With Community-Based Lifestyle Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Smart Aging Program
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Aging; Health Behavior
Keywords: exercise program; lifestyle changes; fitness program; lifestyle intervention
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Aging Program (Experimental): Participants will be enrolled into the Smart Aging Program.
  Interventions: Behavioral: Smart Aging Program
- Control Group (Active Comparator): Participants will be enrolled into group that receives educational materials that reflect the current standard of care.
  Interventions: Behavioral: Educational Materials

INTERVENTIONS:
Behavioral: Smart Aging Program — Comprehensive lifestyle and fitness program designed to improve the health of older adults. The Smart Aging Program represents a package consisting of a dedicated health coach, mobile monitoring, specialized curriculum, and exercise opportunities.
  Arms: Smart Aging Program
Behavioral: Educational Materials — Current standard of care. Includes education materials covering benefits of a healthy lifestyle.
  Arms: Control Group

SUMMARY:
The purpose of this study is to test the efficacy of delivering an exercise and healthy lifestyle program, Smart Aging, to older adults.

DETAILED DESCRIPTION:
The Smart Aging Program is designed to be scalable, implementable, and sustainable in the real world. This program joins patients and their clinicians with community-based fitness centers. The Smart Aging Program looks to use already existing resources to deliver an innovative program to increase physical activity in older adults.

The program begins at the patient-physician level. The program is conducted in community-based fitness centers, the participant's home (home exercise, monitoring) and also sends physical activity data back to the clinician using mobile technology.

The Smart Aging Program consists of a personalized and structured exercise program combined with lifestyle education and mobile-health monitoring. The exercise program includes a 12-week initiation phase, followed by a 40-week maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Clinician referred
* Ambulatory: walk unassisted and successfully complete the 6 minute walk test without rest
* Sufficiently fluent in English to participate in study procedures
* Sedentary or underactive by the Telephone Assessment of Physical Activity61

Exclusion Criteria:

* Clinically-significant systemic or psychiatric illness that may affect safety or completion
* Diagnosis of dementia; use of dementia medications (cholinesterase inhibitors, memantine)
* Myocardial infarction or unstable coronary artery disease (e.g., angina, arrhythmia) in last 6 months.
* Cerebrovascular event (stroke or transient ischemic attack) in the last 6 months
* Cancer diagnosis in the last 2 years (except non-metastatic basal or squamous cell carcinoma or cancer in remission in the absence of treatment for at least 2 years)
* Significant pain or musculoskeletal disorder limiting the ability to participate safely
* Another member of the household enrolled in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 219 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness | Change from Baseline to 12 Weeks
  Measured by peak oxygen consumption (VO2 peak) during treadmill testing.
Change in Cardiorespiratory Fitness | Change from Baseline to 52 Weeks
  Measured by peak oxygen consumption (VO2 peak) during treadmill testing.

SECONDARY OUTCOMES:
Changes in Insulin Resistance | 52 Weeks
  Measured using Homeostasis Model Assessment 2.
Change in Fat Mass | 52 Weeks
  Measured using a dual energy x-ray absorptiometry (DEXA) scan.
Change in Lean Mass | 52 Weeks
  Measured using a dual energy x-ray absorptiometry (DEXA) scan.
Change in Cholesterol | 52 Weeks
  Changes in total cholesterol, LDL, and HDL will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Burns, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Holden R, Szabo-Reed AN, Watts A, Clutton J, Finley K, Wolff SF, Burns JM. Physician referral is associated with recruitment, motivation, and adherence in an exercise intervention study for older adults. J Natl Med Assoc. 2025 Nov 15:S0027-9684(25)00342-6. doi: 10.1016/j.jnma.2025.11.002. Online ahead of print. PMID 41298205
- [Derived] Watts A, Szabo-Reed A, Baker J, Morris JK, Vacek J, Clutton J, Mahnken J, Key MN, Vidoni ED, Burns JM. LEAP! Rx: A randomized trial of a pragmatic approach to lifestyle medicine. Alzheimers Dement. 2024 Dec;20(12):8374-8386. doi: 10.1002/alz.14265. Epub 2024 Oct 8. PMID 39376152